CLINICAL TRIAL: NCT02362399
Title: Effect of Sildenafil Citrate on Uteri- Placental Perfusion, Doppler Indices in Growth Restricted Fetuses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Hayat National Hospital (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: menoufia ob/gyn 1
Record Dates: First submitted 2015-02-05; First posted 2015-02-12 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Pregnancy Complication
MeSH Terms: conditions — Pregnancy Complications | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sildenafil citrate (Active Comparator): 50 mg single oral dose
  Interventions: Drug: sildenafil citrate
- placebo (Active Comparator): single tablet of placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: sildenafil citrate — single oral dose of 50 mg
  Arms: sildenafil citrate
Other: placebo — single oral dose of placebo tablet
  Arms: placebo

SUMMARY:
To detect the effect of sildenafil citrate on Doppler parameters in fetuses suffering from growth restriction to support its use later as prolonged therapy in those pregnancies at higher risk for such complication.

DETAILED DESCRIPTION:
Participants were randomized in 1:1 ratio into one of the following drug regime:

Group (I): "sildenafil citrate group" This group consisted of 22 women who received single oral dose of 50 mg sildenafil citrate.

Group (II): "placebo group" This group consisted of 22 women who received single oral dose of placebo. All participants were evaluated by ultrasound once they admitted and again after 2-hours following administration of either of the treatment tablets. One sonographer was allocated to evaluate all mothers included in the study.

ELIGIBILITY:
Inclusion Criteria:

Patients were admitted to the study based on the following inclusion criteria:

1. Any age and any party.
2. Body mass index between 25 and 35.
3. Singleton pregnancy.
4. Gestational age of 24 weeks or more. Gestational age was established on the basis of menstrual dates and confirmed by first or second trimester ultrasound for booked patients, however, if a difference of > 7 days or > 10 days during first or second trimester respectively, then ultrasound value was used. For unbooked patients they still have the chance to be included in our study if they can bring a scan that showed gestational age during the same period mentioned before.
5. Idiopathic intrauterine growth restriction.
6. Intrauterine growth restriction due to maternal malnutrition, maternal medical disorder as anemia, pregnancy induced hypertension, or chronic renal disease.
7. Intrauterine growth restriction due to substance abuse (including smoking).
8. With or without past history of intrauterine growth restriction .

Exclusion Criteria:

1. Intrauterine growth restriction due to fetal causes as congenital abnormalities, fetal infection, or multiple gestation.
2. Any drug therapy that can affect fetal growth or fetal blood supply.
3. Maternal diseases that contraindicates the use of sildenafil citrate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
improvement of the Doppler indices following treatment | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Shebin Elkom, Egypt

REFERENCES:
- [Derived] El-Sayed MA, Saleh SA, Maher MA, Khidre AM. Utero-placental perfusion Doppler indices in growth restricted fetuses: effect of sildenafil citrate. J Matern Fetal Neonatal Med. 2018 Apr;31(8):1045-1050. doi: 10.1080/14767058.2017.1306509. Epub 2017 Mar 27. PMID 28345432